CLINICAL TRIAL: NCT03343028
Title: Biomarker Establishment for Superior Treatment of PTSD
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: New Mexico VA Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Alan Schatzberg, Kenneth T. Norris, Jr. Professor of Psychiatry and Behavioral Sciences, Stanford University
Other Study IDs: 39006
Record Dates: First submitted 2016-11-04; First posted 2017-11-17 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: PTSD
Keywords: veterans; post traumatic stress disorder; depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Psychotherapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Psychotherapy: The investigators will assess and acquire data on these Veterans across the course of the project prior to and after receiving Prolonged Exposure (PE) or Cognitive Processing Theory (CPT) treatment at VA Palo Alto (VAPAHCS) and the Albuquerque VA. They will acquire fMRI, behavioral, EEG, TMS/EEG, and saliva at baseline on these Veterans and again 3 months after treatment to assess prediction and durability of the clinical and brain/behavioral metrics. All study assessments will take place at Stanford University/VAPAHCS. Subjects will be recruited through VAPAHCS and Albuquerque VA. Subjects will complete a clinical assessment including: neuroimaging, self-report questionnaires completed via computer or paper-and-pencil, cognitive testing, saliva, and TMS and EEG assessments.
  Interventions: Other: Psychotherapy
- Healthy Controls: The investigators will assess and acquire data on these Veterans who do not have history of PTSD and have no history of any Axis I psychiatric disorder, are taking psychotropic medication, or use illicit drugs. They will acquire fMRI, behavioral, EEG, TMS/EEG, and saliva once. All study assessments will take place at Stanford University. Subjects will be recruited through public flying, online ads and VAPAHCS. Subjects will complete a clinical assessment including: neuroimaging, self-report questionnaires completed via computer or paper-and-pencil, cognitive testing, saliva, and TMS and EEG assessments.

INTERVENTIONS:
Other: Psychotherapy
  Other Names: Cognitive Processing Therapy; Prolonged Exposure
  Groups: Psychotherapy

SUMMARY:
The purpose of Biomarker Establishment for Superior Treatment of PTSD is to accelerate research on the discovery of biological, neurological and neuroimaging markers for Post- Traumatic Stress Disorder (PTSD). The investigators hope to validate and extend the network efficiency and verbal memory biomarker for PTSD. The investigators hope to learn whether there are pretreatment biological factors that can predict response to therapy. They want to do this by understanding the brain network function, relating EEG to functional magnetic resonance imaging, and application of network analysis tool.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD by VA clinicians and acceptance into PE or CPT treatment as part of the PCT
* Veterans of any era

Exclusion Criteria:

* MRI safety contraindications
* Active, uncontrolled medical illness
* Acute suicidality
* Current substance dependence
* Current use of thyroid medication or active hyper/hypothyroidism
* Neurological disorder affecting the CNS Seg stroke, epilepsy, tumorW or penetrating head injury
* Use of PRN within 48 hours of the MRI/EEG

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: We will assess and acquire data on these Veterans across the course of the project prior to and after receiving Prolonged Exposure (PE) or Cognitive Processing Theory (CPT) treatment at VA Palo Alto (VAPAHCS) and the Albuquerque VA.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2016-09; Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Understanding the brain network function-neuroimaging and behavioral with Clinician-Administered PTSD Scale for DSM-5 | Approximately 3 months
  We will be using CAPS 5

CONTACTS AND LOCATIONS:
Overall Officials: Alan Schatzberg, MD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - VA Palo Alto Health Care System (VAPAHCS), Palo Alto, California
  - New Mexico VA Health Care System, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No